CLINICAL TRIAL: NCT03609619
Title: A Multicenter, 2-Part, 6-Week, Double-blind, Randomized, Placebo-controlled, Parallel-design Study to Assess the Efficacy and Safety of AEVI-001 in Children and Adolescents (Ages 6-17 Years) With Attention Deficit Hyperactivity Disorder and With or Without Copy Number Variants in Specific Genes Implicated in Glutamatergic Signaling and Neuronal Connectivity
Brief Title: PART B: Efficacy and Safety of AEVI-001 in Children and Adolescents With ADHD and Without mGluR Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Responsible Party: Sponsor
Organization: Avalo Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEVI-001-ADHD-202B
Record Dates: First submitted 2018-07-31; First posted 2018-08-01 (Actual); Results first posted 2019-07-16 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2019-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AEVI-001 (Experimental)
  Interventions: Drug: AEVI-001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AEVI-001 — Oral doses of 100 mg, 200 mg or 400 mg of AEVI-001 will be administered twice daily, during the treatment period.
  Other Names: MDGN-001; NFC-1
  Arms: AEVI-001
Drug: Placebo — Oral doses of Placebo will be administered twice daily, during the treatment period.
  Arms: Placebo

SUMMARY:
This is PART B of a 2-part, 6-week, double-blind, dose-optimization, parallel-group study in children and adolescents (ages 6-17 years) with ADHD with and without CNVs in specific genes implicated in glutamatergic signaling and neuronal activity. PART B will assess subjects who do not have CNVs in any of the specific gene mutation(s) implicated in glutamatergic signaling and neuronal connectivity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject and parent/legally authorized representative (LAR) can speak English fluently and have provided written informed consent, and assent (as applicable) for this study.
2. Subject is 6 to 17 years of age (inclusive) at the time of consent/assent. The date of signature of the informed consent/assent is defined as the beginning of the Screening Period. This inclusion criterion will only be assessed at the Screening Visit (Visit 1).
3. Subject is male or non-pregnant, non-lactating female, who if of childbearing potential agrees to comply with any applicable contraceptive requirements prior to administration of investigational product (IP).
4. Subject meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD based upon DSM 5 criteria.
5. Subject has a minimum score of ≥28 on the ADHD-RS-5 at the Baseline Visit (Visit 2).
6. Subject has been genotyped previously and has their identity confirmed (if required).

Exclusion Criteria:

1. Subject or parent/LAR is, in the opinion of the investigator, mentally or legally incapacitated, has significant emotional problems at the time of the Screening Visit (Visit 1) which could interfere with the conduct of study evaluations.
2. Subject has a current, controlled or uncontrolled, co-morbid major psychiatric diagnosis (aside from ADHD), including an anxiety disorder, major depression, bipolar disease, schizophrenia (or any psychotic disorder), and moderate or severe intellectual disability. Mild anxiety and/or depressive symptoms that do not meet diagnostic criteria for an anxiety disorder or major depression and/or do not require treatment are not exclusionary.
3. Subject has autism spectrum disorder to include a DSM-IV diagnosis of autistic disorder, Asperger's disorder, or pervasive developmental disorder.
4. Subject is currently taking any medication that might confound the results of safety assessments conducted in the study.
5. Subject has a known history of cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, cardiac conduction problems, exercise-related cardiac events including syncope and pre-syncope, or other serious cardiac problems.
6. Subject has any clinically significant abnormality on 12-lead ECG performed at the Screening Visit (Visit 1) and/or the Baseline Visit (Visit 2) such as serious arrhythmia, cardiac conduction problems, or other abnormalities deemed to be a potential safety issue.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aevi Genomic Medicine, Wayne, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AEVI-001: Oral doses of 100 mg, 200 mg or 400 mg administered b.i.d.
- Placebo: Oral doses of Placebo administered b.i.d.
Period: Overall Study
Arm/Group | AEVI-001 | Placebo
Started | 54 | 55
Completed | 44 | 49
Not Completed | 10 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 2
Not completed — Protocol Violation | 5 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: ITT Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | AEVI-001 | Placebo | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (3.04) | 10.3 (2.70) | 10.4 (2.86)
Age, Customized [Count of Participants; unit: Participants]
  6 to 12 years | 41 | 42 | 83
  13 to 17 years | 12 | 13 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 34 | 36 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 20
  Not Hispanic or Latino | 41 | 46 | 87
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 41 | 41 | 82
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 53 | 55 | 108
Attention Deficit Hyperactivity Disorder Rating Scale, Version 5 (ADHD-RS-5) Total Score [Mean (Standard Deviation); unit: units on a scale] — The ADHD-RS-5 is comprised of 18 frequency items and 12 impairment items. Each frequency item was scored on a scale from 0 = "Never or rarely" to 3 = "Very often".
  The ADHD-RS-5 total score was calculated as the sum of the 18 frequency item scores. The total score ranges from 0 to 54. Higher scores indicate greater symptom severity.
  units on a scale | 40.5 (8.78) | 40.6 (8.71) | 40.6 (8.70)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale, Version 5 (ADHD-RS-5) Total Score
Description: The ADHD-RS-5 is comprised of 18 frequency items and 12 impairment items. Each frequency item was scored on a scale from 0 = "Never or rarely" to 3 = "Very often".
  The ADHD-RS-5 total score was calculated as the sum of the 18 frequency item scores. The total score ranges from 0 to 54. Higher scores indicate greater symptom severity. Change from baseline value were calculated as the assessment value minus the baseline value.
Time Frame: Baseline to Visit 8 (Week 6)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AEVI-001 | Placebo
Number analyzed (Participants) | 52 | 54
units on a scale | -11.04 (1.730) | -10.38 (1.651)

2. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI -I) Response
Description: The CGI-I item is rated on a 7-point scale from 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", 7 = "Very much worse".
  Response is defined as achieving a CGI-I score of 1 or 2, scores of 3 to 7 or missing are defined as Non Response
Time Frame: Visit 3 to Visit 8 (Week 6)
Measure: Count of Participants; unit: Participants
Arm/Group | AEVI-001 | Placebo
Number analyzed (Participants) | 52 | 54
Participants | 15 | 16

ADVERSE EVENTS:
Time Frame: 3 months, 13 days
Description: All AEs are collected from the time of the informed consent is signed until the follow-up call is completed. This includes events occurring during the screening phase of the study, regardless of whether investigational product (IP) is administered. An AE will be considered treatment emergent if it occurs after the first dose of IP and within 3 days of a subjects last dose of IP.
Arm/Group | AEVI-001 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/55
Other Adverse Events (participants affected / at risk) | 3/53 | 9/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AEVI-001 (N=53) | Placebo (N=53)
Weight increased (Investigations) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 3 (6) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The information generated by this study is the property of Aevi Genomic Medicine, Inc. Publication or other public presentation of AEVI-001 data resulting from this study requires prior review and written approval of Aevi Genomic Medicine, Inc. Abstracts, manuscripts, and presentation materials should be provided to Aevi Genomic Medicine, Inc. for review at least 30 days prior to the relevant submission deadline.

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT03609619/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03609619/SAP_001.pdf